CLINICAL TRIAL: NCT02835586
Title: STREAMER : Stent Restenosis and Medicaments Release : Does Local Delivery of Paclitaxel be Safe and Efficient in Stenting of TransAtlantic InterSociety Consensus (TASC) Class C and D Femoropopliteal Artery Lesions
Brief Title: STREAMER : STent Restenosis And MEdicaments Release
Acronym: STREAMER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-701
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Critical Ischemia
Keywords: paclitaxel; critical ischemia; restenosis; femoropopliteal artery lesions TASC C and D
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paclitaxel delivery in femoropopliteal artery (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel will be administered intra-arterially through an irrigating catheter to treat a diseased segment of superficial femoral artery and/or popliteal artery after stenting. Dosing will be based on the lesion surface area and will be calculated using the following formula : 22/7 x diameter (mm) x length (mm) x 3 µg/mm3

SUMMARY:
It is a pilot study to evaluate the feasibility and the efficiency of local delivery of paclitaxel after stenting of long femoropopliteal arterial lesions TASC C and D before the realization of a large randomized multicentric study. Patients concerned are in critical ischemia.

ELIGIBILITY:
Inclusion Criteria:

* patients with critical ischemia of a lower limb with ankle pressure < 50 mmHg
* lesions TASC C and D of the superficial femoral or popliteal artery

Exclusion Criteria:

* patient allergic to paclitaxel
* patient with a cancer, a neutropenia, with immunosuppressor medicament or chemotherapy
* patient with contraindication to take 2 anti-aggregants platelets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with femoropopliteal artery restenosis | 12 months
  defined as restenosis > 50 % with a velocity pick > 2,5 on duplex ultrasound

SECONDARY OUTCOMES:
Occurence of adverse events due to paclitaxel | From1 day to 12 months
  biological adverse events (thrombopenia, neutropenia)
Number of patients with target lesion revascularization | 12 months
  number of subjects who need a new revascularization on the same artery (femoropopliteal)
Occurence of amputation free-survival | 12 months
cumulated rate of morbi-mortality (TCMM) | up to 30 days
  myocardial infarction, death, vascular ischemic accident, cardiac angina, major amputation, new hospitalization or new surgery for hematoma, thrombosis or false aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Nellie DELLA SCHIAVA, MD, Principal Investigator — department of vascular surgery, Edouard Herriot Hospital, LYON
Locations (1):
- department of vascular surgery, Edouard Herriot Hospital, 5 Place d'Arsonval, Lyon, France